CLINICAL TRIAL: NCT06601049
Title: Effectiveness of ResArgin on Adult's Body Composition and Health: a Randomized Double-Blind Placebo-Controlled Trial
Brief Title: Effectiveness of ResArgin on Adult's Body Composition and Health
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Heather Hausenblaus (Other)
Responsible Party: Sponsor-Investigator, Dr. Heather Hausenblaus, Professor, Jacksonville University
Organization: Jacksonville University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WDL022024
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ResArgin (Active Comparator): A resveratrol-based supplement. Participants will receive a daily oral dose of ResArgin containing [50 mg/d] of trans-Resveratrol for 90 days.
  Interventions: Dietary Supplement: ResArgin
- placebo (Placebo Comparator): Placebo consists of oat hull. Participants receive a daily oral dose of a placebo matching the appearance and dosage form of ResArgin for 90 days.
  Interventions: Dietary Supplement: ResArgin

INTERVENTIONS:
Dietary Supplement: ResArgin — Resveratrol-based supplement

SUMMARY:
The goal of this clinical trial is to learn if the supplement ResArgin (a reservatrol-based supplement) works to slow down muscle loss during a period of fat loss. Other related health outcomes such as sleep, mood, and activity will be assessed. The main questions it aims to answer are:

Does ResArgin improve muscle loss? Does ResArgin improve sleep quality, activity, mood, and body satisfaction.

Researchers will compare ResArgin to a placebo (a look-alike substance that contains no active ingredients) to see if ResArgin works to improve muscle loss and related health outcomes.

Participants will:

Take ResArgin or the Placebo every day for 3 months

Assessment will occur at Baseline, Day 30, Day 60, and Day 90.

Participants will complete a daily diary of their mood and health.

DETAILED DESCRIPTION:
Study Purpose: Examine the effectiveness of ResArgin in attenuating muscle loss during a period of fat loss in overweight and mildly obese men and women.

Outcomes: Primary outcomes will be body composition. Secondary outcomes will be physical activity, food cravings, health-related quality of life, body satisfaction, basal metabolic rate, sleep behaviors, mood, anxiety, and perceived stress.

Study Design • Randomized double-blind placebo-controlled trial

o N = 60 men and women (30 adults in the ResArgin Condition and 30 adults in the Placebo Condition).

ELIGIBILITY:
Inclusion Criteria:

* overweight and mildly obese adults
* age range between 25 to 60 years

Exclusion Criteria:

* metabolic or endocrine related dysregulation including but not limited to: diagnosis of type I or type II diabetes, liver, kidney, or pancreatic dysfunction.
* history of seizures or epilepsy-related disorders
* musculoskeletal issues that would prohibit them from engaging in spontaneous activity,
* metabolic disorder
* sleep disorder
* psychiatric condition
* dietary aversions or restrictions including any animal sources of protein, dairy, fruits/vegetables, nut/seed allergy, eggs, and wheat/gluten or are currently following a carbohydrate restricted (under 20%) habitual diet.
* smokers
* consume excessive amounts of alcohol (>3 drinks/d)
* actively intermittent fasting
* actively trying to lose weight or have lost more than ± 3kg in previous 3 months
* pregnant
* nursing
* trying to conceive
* changed their birth control in the past 3 months.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Body composition change from baseline in fat mass and fat free mass as assessed by a DEXA scan at 90 days | From enrollment to the end of intervention at 90 days
  This will be assessed objectively by a trained health professional.

SECONDARY OUTCOMES:
Change from baseline in health-related quality of life, sleep quality, activity, and mood at 90 days | Change from Baseline to Day 90
  Health-related quality of life where zero is equivalent to high quality of life and 30 indicates the worst quality of life. Sleep quality as assessed by the Insomnia Severity Index where 0 indicates excellent sleep quality and 28 indicates worst sleep quality. Mood as assessed by the Profile of Mood States where 0 = Not at all and 4 = Extremely. Sleep quality and activity as assessed by the Oura Ring where 0 indicates poor sleep quality or activity and 100 indicates excellent sleep quality and activity. Bioelectrical impedance scale assessed percent body fat where a higher score indicates a higher percent body fat.

CONTACTS AND LOCATIONS:
Locations (1):
- Jacksonville University, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Gateway Health Alliance will determine the IPD sharing plan